CLINICAL TRIAL: NCT00926744
Title: Large-Scale Randomized Intervention Trial of Effects of Physical Activity on Incidence and Risk Factors of Cardiovascular Diseases in Healthy People
Brief Title: Nutrition and Exercise Intervention Study
Acronym: NEXIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Motohiko Miyachi, Chief, Department of Health Promotion and Exercise, National Institute of Health and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: qde402mm; 21170901
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Dyslipidemia; Diabetes; Low Back Pain
Keywords: physical activity; nutrition; cardiovascular diseases; musculo-skeletal problems
MeSH Terms: conditions — Hypertension; Dyslipidemias; Diabetes Mellitus; Low Back Pain; Motor Activity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention (Experimental): Physically inactive participants receiving both physical activity and dietary counseling
  Interventions: Behavioral: physical activity
- Active (No Intervention): Physically active participants receiving only dietary counseling
- Control (No Intervention): Physically inactive participants receiving only dietary counseling

INTERVENTIONS:
Behavioral: physical activity — The targets of amount of physical activity are 3.3METs•h/day (MVPA) and 10,000 step counts/day.
  Arms: Intervention

SUMMARY:
The purpose of the present study was to clarify the effects of increase in physical activity on incidence and surrogate marker of cardiovascular diseases. The working hypothesis of the present study was that the physical activity to satisfy the Japanese guideline of Ministry of Health, Labour and Welfare is effective for the primary prevention of the lifestyle-related disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 30-64 years old

Exclusion Criteria:

* During treatment of any diseases
* Two or more metabolic risk factors

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1085 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Objectively measured amount of physical activity | 10 years

SECONDARY OUTCOMES:
Surrogate measurement of lifestyle-related diseases (blood pressure, FPG, cho, etc) | 5 years
Incidence of lifestyle-related diseases (hypertension, dyslipidemia, diabetes) | 10 years
Incidence of musculoskeletal and joint pain | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Health and Nutrition, Shinjuku, Tokyo, Japan

REFERENCES:
- [Derived] Tripette J, Gando Y, Murakami H, Kawakami R, Tanisawa K, Ohno H, Konishi K, Tanimoto M, Tanaka N, Kawano H, Yamamoto K, Morishita A, Iemitsu M, Sanada K, Miyatake N, Miyachi M. Effect of a 1-year intervention comprising brief counselling sessions and low-dose physical activity recommendations in Japanese adults, and retention of the effect at 2 years: a randomized trial. BMC Sports Sci Med Rehabil. 2021 Oct 25;13(1):133. doi: 10.1186/s13102-021-00360-7. PMID 34696811